CLINICAL TRIAL: NCT00842595
Title: Phase II Study of Treatment of Relapsed Agressive Lymphomas
Brief Title: Efficacy , Safety of Treatment R NIMP for Relapsed Aggressive Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R NIMP
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2010-07

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: relapsed aggressive B-cell lymphoma; Chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Vinorelbine; Ifosfamide; Mitoxantrone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R NIMP (Experimental): (Mabthera®) Rituximab IV 375 mg/m²day 1 (Navelbine ®)Vinorelbine IV 25mg/m² day 1 and day 5 (Novantrone®)Mitoxantrone IV 10 mg/m² day 1 (Holoxan®)Ifostamide IV 1000 mg/m²day 1 to day 5 (Cortancyl®)prednisone oral day 1 to day 5
  Interventions: Drug: rituximab; Drug: vinorelbine; Drug: ifosfamide; Drug: Mitoxantrone; Drug: Prednisone

INTERVENTIONS:
Drug: rituximab — 6 courses every 28 days
  Other Names: (Mabthera ® )Rituximab IV 375 mg/m²day
Drug: vinorelbine — 6 courses every 28 days
  Other Names: (Navelbine ®) Vinorelbine IV 25mg/m² day 1 and day 5
Drug: ifosfamide — 6 courses every 28 days
  Other Names: (Holoxan®)Ifostamide 1000mg/m² day 1 to day 5
Drug: Mitoxantrone — 6 courses every 28 days
  Other Names: (Novantrone®) Mitoxantrone 10mg/m² day1
Drug: Prednisone — 6 courses every 28 days
  Other Names: (Cortancyl®)Prednisone 1m/kg day 1 to day 5

SUMMARY:
The primary objective of the protocol is to estimate the complete response rate of three courses of the association of rituximab, navelbine, ifosfamide, mitoxantrone, and prednisone in relapsed aggressive non hodgkin's B-cell lymphoma

DETAILED DESCRIPTION:
Phase II study of the efficacy and toxicity of rituximab, navelbine, ifosfamide, mitoxantrone, and prednisone in relapsed aggressive non hodgkin's B-cell lymphoma.

The study intervention is an administration of 3 courses of the abovementioned drugs, witch doses are detailed below. Remission is assessed and the investigator is free to proceed with any kind of consolidation , he decides best for the patient( high dose or standard chemotherapy).

The addition of Rituximab the the NIMP protocol is warranted on the basis of previous publications wtich have shown a significant advantage in addition to chemotherapy in complete remission rate and in overall survival.

Navelbine has shown an interesting activity in lymphoma relapse. Mitoxantrone has a good toxicity profile for patients who have prevously received anthracyclines, and there is not so much cross resistance between the two drugs.

Ifosfamide is commonly used in the treatment of relapsed and refractory lymphoma, because of its low hematologic toxicity profile and good antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, between 18 and 75 years old
* CD 20+ large cell lymphoma
* In first relapse
* No previous autologous stem cell transplantation or relapsing more than 12 months after an autologous stem cell transplantation
* Ann Arbor stage I, II, III ou IV
* ECOG 0,1 or 2
* Signed informed consent

Exclusion Criteria:

* age: before 18 and more than 75 years old
* other type of lymphoma
* Informed consent not signed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-12; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Complete remission rate | CR AFTER 3 R NIMP COURSES

SECONDARY OUTCOMES:
overall remission rate | OS after 3 R NIMP COURSES
Toxicity | R NIMP TOLERANCE
Pharmacoeconomy | treatment phramacoeconomy

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel GYAN, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Hôpital COCHIN, Paris, France